CLINICAL TRIAL: NCT00246948
Title: The Efficacy of Active Conservative Treatment for Patients With Severe Sciatica. A Randomized Clinical Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Back Research Center, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VF 20010134
Record Dates: First submitted 2005-10-31; First posted 2005-11-01 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2005-10

CONDITIONS: Sciatica
Keywords: Physical therapy
MeSH Terms: conditions — Sciatica

INTERVENTIONS:
Procedure: Active conservative treatment of sciatica

SUMMARY:
This Study si designed as a Prospective clinical controlled randomized trial.

Background:

Reviews have demonstrated no or little efficacy for passive conservative treatment modalities for patients suffering from sciatica. The results of surgery are conflicting. Cohort studies have shown a high efficacy for active treatment modalities in patients with sciatica. The current trend in treatment of low back pain without sciatica is focusing on active conservative treatment like information and advice to stay active and exercises.

Aim: To evaluate the efficacy of two active conservative treatment programs for patients with severe sciatica.

Methods: In a prospective clinical controlled randomized trial, 181 consecutive patients with radicular pain below the knee were examined at baseline, 8 weeks later at post treatment follow-up, and at one year follow-up and MR-scanned at baseline and one year follow-up. The treatment consisted of four elements: 1-3 were identical in both groups. 1. Thorough information concerning anatomy, pathogenesis, how discs heal without surgery, and encouragement to stay as active as possible but to reduce activity if an increase in leg pain occurs. 2." Tender love and care". 3. Medication; this was optional and only weak analgesic and NSAIDs were recommended.

Element 4 consisted of two different exercise programs. Symptom guided exercises consisted of a variety of back related exercises and optional manual treatment. The exercises were given after an algorithm, where different symptoms or a response to exercises determined the exercises given. The other group, Sham exercises had voluntary not back related exercises. The exercises were aimed at increasing the general blood circulation and maintaining strength in the extremities. Outcome measures were functional status, pain, MRI findings, clinical findings, and history

DETAILED DESCRIPTION:
Summary of Background Data. Sciatica as a result of a herniated disk is a fairly common problem; studies have shown a life time prevalence of 4-5 % in the Scandinavian population. Though a herniated disk is a benign disease with a relatively good prognosis, the pain and functional loss, are in most patients rather considerable over a period of some months Reviews have demonstrated no or little efficacy for passive conservative treatment modalities. Results for surgery are conflicting. Cohort studies have shown a high efficacy for active treatment modalities in patients with sciatica.

The current trend in back treatment is information and advice to stay active including active treatment modalities in which patients are given responsibility during the treatment process and the treatment assumes the role of a "coach".

Objectives. To evaluate the efficacy of two active conservative treatment programs for patients with severe sciatica.

Methods A prospective clinical controlled randomized trial including 181 consecutive patients with radicular pain below the knee. The patients were examined at baseline, 8 weeks later at post treatment follow-up, and, and MR-scanned at baseline and at the one year follow-up The treatment consisted of four elements; 1-3 were identical in both groups. 1. Thorough information concerning anatomy, pathogenesis, how discs heal without surgery, and encouragement to stay as active as possible but to reduce activity if an increase in leg pain occurs. 2. Tender love and care. 3. Medication, this was optional and only weak analgesic and NSAID'S were recommended.

Element 4 was divided into a "Hands on" and "Hands off", utilizing two different exercise programs. "Hands on" consisted of a variety of back related exercises and optional manual treatment. The exercises were given after a strict algorithm, where different symptoms or a response to exercises determined the exercises given.

"Hands off" exercises were optional and generally not back related. They were geared towards increasing general blood circulation and maintaining strength in the extremities.

ELIGIBILITY:
Inclusion Criteria:

* Radicular pain of dermatonal nature in one or both legs or below the knee Leg pain > 3 on the eleven point box scale20 Radiating pain duration between two weeks and one year Age between 18 to 65 years

Exclusion Criteria:

- Cauda equine syndrome Not having Danish as first language Pending workers litigation claims Inability to follow the rehabilitation protocol, due to concomitant disease Previous back surgery Spinal tumors Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181
Dates: Start 2001-11; Study Completion 2003-08

CONTACTS AND LOCATIONS:
Overall Officials: Hanne B Albert, Ph.D., Principal Investigator — The Back Research Center, Funen
Locations (1):
- The Back Research Center, Ringe, Denmark